CLINICAL TRIAL: NCT07305519
Title: The Combined Effect of Magnesium, Palmitoylethanolamide, High-Molecular-weight Hyaluronic Acid, Vitamin B6, and Vitamin D in Preventing Preterm Birth: A Randomized Controlled Trial
Brief Title: The Combined Effect of Magnesium, Palmitoylethanolamide, High-Molecular-weight Hyaluronic Acid, Vitamin B6, and Vitamin D in Preventing Preterm Birth:
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Rizzo, Prof. Giuseppe Rizzo, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEATB_2025
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Preterm Labor
Keywords: preterm labor; preterm birth; prematurity; magnesium; hyaluronic acid; vitamin B6; Vitamin D
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: Magnesium-PEA-HMW Hyaluronic Acid-Vitamin B6-Vitamin D + Vaginal Progesterone (Experimental)
  Interventions: Drug: Magnesium-PEA-HMW Hyaluronic Acid-Vitamin B6-Vitamin D + Vaginal Progesterone
- Control: Vaginal Progesterone Only (Active Comparator)
  Interventions: Other: Standard Treatment (Guideline-Based)

INTERVENTIONS:
Drug: Magnesium-PEA-HMW Hyaluronic Acid-Vitamin B6-Vitamin D + Vaginal Progesterone — Participants randomized to the treatment arm will receive a combination oral supplement containing Magnesium (450 mg), Palmitoylethanolamide (200 mg), high-molecular-weight Hyaluronic Acid (200 mg), Vitamin B6 (2.6 mg), and Vitamin D (50 µg / 2000 IU), administered as two tablets per day. The supplement will be given in addition to standard vaginal progesterone (200 mg once daily). Treatment begins at enrollment (20-34 weeks' gestation) and continues until 37 weeks of gestati
  Arms: Treatment: Magnesium-PEA-HMW Hyaluronic Acid-Vitamin B6-Vitamin D + Vaginal Progesterone
Other: Standard Treatment (Guideline-Based) — Participants randomized to the control arm will receive standard therapy consisting of vaginal progesterone (200 mg once daily) from enrollment (20-34 weeks' gestation) until 37 weeks of gestation. No additional supplements or investigational products will be administered.
  Arms: Control: Vaginal Progesterone Only

SUMMARY:
The aim of the study is to assess the effect of a combination of Magnesium, Palmitoylethanolamide, high-molecular-weight Hyaluronic Acid, Vitamin B6, and Vitamin D in women at risk of preterm birth (PTB).

DETAILED DESCRIPTION:
Preterm birth (PTB) remains one of the leading causes of neonatal morbidity and mortality worldwide. The transition of the myometrium from a quiescent state to active contractility is driven by a complex interplay of genetic predisposition, inflammatory mediators, endocrine factors, and uterine environmental conditions. Increased expression of pro-inflammatory cytokines (including IL-6, IL-1β, TNF-α), activation of NF-κB pathways, prostaglandin synthesis, cervical remodeling, and alterations in progesterone signaling contribute to the premature onset of labor.

Several natural molecules have demonstrated potential roles in modulating uterine quiescence, inflammatory pathways, and cervical integrity. Magnesium participates in more than 600 enzymatic reactions and reduces inflammatory cytokine production, while low serum magnesium levels have been associated with a higher risk of PTB. Vitamin B6 contributes to fetal neurodevelopment and has been linked to reduced rates of preeclampsia and preterm birth. High-molecular-weight hyaluronic acid (HMWHA) plays a crucial role in immune tolerance at the maternal-fetal interface, promotes anti-inflammatory cytokine secretion, and supports progesterone-mediated uterine quiescence through upregulation of the progesterone receptor membrane component-1 (PGRMC1). Palmitoylethanolamide (PEA), an endogenous bioactive lipid, exerts anti-inflammatory and mast-cell-stabilizing properties and has been found at significantly higher levels in women with PTB as part of a compensatory physiological response. Vitamin D, a steroid-like hormone, modulates immune pathways and downregulates CRH, prostaglandin production, and oxytocin signaling, all of which are implicated in the initiation of labor.

This randomized, prospective, open-label pilot study aims to evaluate whether the combination of Magnesium, Palmitoylethanolamide, high-molecular-weight Hyaluronic Acid, Vitamin B6, and Vitamin D, administered in addition to standard vaginal progesterone, can reduce the incidence of preterm birth in women at increased risk due to a sonographic cervical length of 15-30 mm between 20 and 34 weeks' gestation.

A total of 150 women with singleton pregnancies will be randomized 1:1 to receive either standard care with vaginal progesterone alone (control group) or vaginal progesterone plus the oral combination supplement (treatment group). Cervical length will be assessed at baseline, 1 week, and 2 weeks after enrollment. Participants will be followed until 37 weeks of gestation or delivery.

The primary outcome is the proportion of women delivering at or beyond 36 weeks of gestation. Secondary outcomes include the incidence of preterm uterine contractions, emergency department visits for uterine contractions, time interval from treatment initiation to delivery, and longitudinal changes in cervical length.

As the first study to investigate this specific molecular association for PTB prevention, it is designed as a pilot trial to generate preliminary efficacy data and inform future larger randomized controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Singleton pregnancy

Maternal age ≥ 18 years

Gestational age between 20+0 and 34+0 weeks at enrollment

Cervical length between 15 mm and 30 mm measured by transvaginal ultrasound

Exclusion Criteria:

* Fetal structural anomalies

Maternal chronic diseases or pregnancy-related conditions, including diabetes, hypertension, preeclampsia, cardiovascular disease, infections, or autoimmune disorders

Multiple gestation

Fetal growth abnormalities (estimated fetal weight <10th or >90th percentile)

Prelabor rupture of membranes (PROM)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Preterm Birth before 37 weeks | Up to 37 weeks of gestation or delivery, whichever occurs first.
  Proportion of participants who deliver before 37+0 weeks of gestation in each study arm.

SECONDARY OUTCOMES:
Incidence of Preterm Uterine Contractions | From enrollment until 37 weeks of gestation or delivery.
  Number of episodes of uterine contractions requiring clinical evaluation, as reported by participants or documented during hospital visits.
Emergency Department Visits for Preterm Contraction | From enrollment until 37 weeks of gestation or delivery.
  Number of emergency department or obstetric triage visits due to symptoms of preterm uterine activity.
Interval From Treatment Initiation to Delivery | From baseline (T0) to delivery.
  Number of days between study enrollment (start of therapy) and delivery.
Change in Cervical Length at 1 Week | Baseline (T0) and 1 week (T1).
  Difference in transvaginal cervical length (mm) between baseline and 1 week after randomization.
Change in Cervical Length at 2 Weeks | Baseline (T0) and 2 weeks (T2).
  Difference in transvaginal cervical length (mm) between baseline and 2 weeks after randomization.

IPD SHARING:
Plan to Share IPD: Undecided